CLINICAL TRIAL: NCT06708663
Title: Phase IIa Study of HX009+IN10018 in Patients with Advanced Solid Tumours, Including Biliary Tract Malignancies and Malignant Melanoma, Treated with or Without Standard Chemotherapy
Brief Title: HX009+ IN10018 with or Without Standard Chemotherapy for Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX009-II-05
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Biliary Tract Cancer; Melanoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HX009+IN10018 (Experimental)
  Interventions: Drug: HX009+IN10018

INTERVENTIONS:
Drug: HX009+IN10018 — The 7.5 mg/kg dose group will first enroll 3 to 6 subjects, and if the 7.5 mg/kg dose group is tolerable, then 3 to 6 subjects will continue to be enrolled into the 10 mg/kg dose group; if the 7.5 mg/kg dose group is not tolerable, a decision will be made to add a new, lower dose group after discussion between the sponsor and the investigator; in addition, based on the available study data, the sponsor and the investigator will discuss and decide whether to add an unplanned dose group or an exploratory group and decide on the appropriate recommended dose (RP2D) for the Phase IIa study.
  IN10018 is fixed dose at 100mg daily.

SUMMARY:
Phase IIa study of HX009+ IN10018 in combination with or without standard chemotherapy in patients with advanced solid tumours including biliary tract malignancies and malignant melanoma

DETAILED DESCRIPTION:
The Part1 safety run-in stage:

About 6~24 patients are expected to be enrolled in the safety run-in stage, 3~6 cases will be enrolled first in the 7.5mg/kg dose group, and if the 7.5mg/kg dose level is tolerable, then 3~6 cases will continue to be enrolled up to the 10mg/kg dose group; if the 7.5mg/kg dose group can not be tolerated, it will be decided whether to add a new lower dose level after discussion between the sponsor and the investigators, based on the '3+3' rule, which determines the actual number of cases enrolled, the number of replacement subjects, and the number of dose groups to be explored for each cohort based on observed safety data.

Part I Phase IIa stage:

Based on data from safety run-in stage , a target ORR of 20% for HX009 in combination with IN10018 in patients with treated advanced biliary cancers was pre-set, and a total of 20-30 subjects were planned to be enrolled at the appropriate recommended dose level, and HX009 in combination with IN10018 for the treatment of patients with advanced biliary malignancies was considered to be a treatment option for HX009 in combination with IN10018 if the best efficacy was observed as a CR or a PR in at least 5 subjects. patients with advanced biliary malignancies, supporting further exploratory studies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the trial and sign the informed consent form;
2. male or female, age at 18 to 70 years (including borderline value) ;
3. expected survival ≥ 12 weeks;
4. ECOG score 0-1;
5. patients with unresectable/metastatic advanced solid tumours (including biliary tract malignancies and malignant melanoma) confirmed by cytology or histopathology; Part I: Failed standard therapy, or no effective standard therapy (prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies may be eligible for enrolment); Part II: No prior systemic therapy (prior neoadjuvant and adjuvant therapy is permitted, but needs to have been completed at least 6 months ago);

Exclusion Criteria:

1. Histological or pathological diagnosis of carcinoma of the jugular abdomen;
2. Patients with melanoma with known BRAF v600E mutation and NRAS mutation; patients with cholangiocarcinoma and gallbladder cancer with known BRAF v600E mutation, NTRK gene fusion, RET gene fusion mutation, FGFR2 gene fusion, IDH1 gene mutation, and KRAS mutation
3. Subjects with symptomatic brain metastases, meningeal metastases, or spinal cord compression, except for the following: asymptomatic brain metastases (i.e., no progressive central nervous system symptoms caused by brain metastases, no need for corticosteroid or antiepileptic drugs, and the lesion has been stable for ≥4 weeks as confirmed by imaging tests);
4. have had a malignancy other than the study disease (biliary malignancy, malignant melanoma) within 5 years prior to signing the ICF, except for malignancies with negligible risk of metastasis or death and/or those that have received curative treatment (e.g. adequately treated cervical carcinoma in situ, basal or squamous cell skin carcinoma, confined prostate cancer, ductal carcinoma in situ, or stage I uterine cancer);
5. Subjects with an active, or history of, autoimmune disease that is likely to recur or is currently being treated (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or at high risk (e.g., organ transplants requiring immunosuppressive therapy). However, subjects with the following diseases were allowed to enrol:

   * Type 1 diabetes mellitus that has stabilised with the use of fixed doses of insulin;
   * Autoimmune hypothyroidism and adrenal insufficiency requiring only hormone replacement therapy;
   * Skin diseases that do not require systemic therapy: e.g. eczema, rashes that cover less than 10 per cent of the body surface, psoriasis without ocular symptoms.
6. have severe cardiovascular disease such as symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina, uncontrolled hypertension (systolic blood pressure ≥160 and/or diastolic blood pressure ≥100 mmHg under pharmacological control), cardiac arrhythmia, history of myocardial infarction within 6 months, or history of arterial thromboembolism or pulmonary embolism within 3 months prior to the first administration of the drug
7. suffering from a serious lung disease requiring treatment or previous serious lung disease, interstitial lung disease, interstitial pneumonitis, pulmonary fibrosis, radiation pneumonitis requiring hormonal therapy, etc;
8. uncontrolled concomitant medical conditions including, but not limited to, severe diabetes mellitus (fasting blood glucose > 250 mg/dl or 13.9 mmol/L), active infectious diseases, psychiatric disorders (e.g., epilepsy) that may interfere with adherence, or other serious conditions requiring systemic therapy
9. patient with uncontrolled pleural effusions, abdominal effusions or pericardial effusions that require repeated drainage. Individuals with indwelling drains are permitted to be enrolled;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
RP2D | Approximately 2 year
  recommended phase 2 dose for HX009 in combination with IN10018 in advanced solid tumor
ORR | approximately 2 years
  objective reponse rate per investigator by RECIST1.1

SECONDARY OUTCOMES:
AEs | approximately 2 years
  occurrency of AEs
PFS | approximately 2 years
  median progress-free survival per RECIST 1.1 by Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China